CLINICAL TRIAL: NCT07000370
Title: Bridging Generations: Educating Children on Dementia and Fall Prevention Through Animation
Acronym: fall
Status: Completed | Type: Observational
Sponsor: Northumbria University (Other)
Responsible Party: Sponsor
Other Study IDs: Animated HomeHazard Assessment
Record Dates: First submitted 2025-05-30; First posted 2025-06-02 (Actual); Last update posted 2025-06-02 (Actual); Status verified 2025-05

CONDITIONS: Fall Prevention in Healthy Aging
Keywords: fall

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Animation: education

SUMMARY:
A retrospective data review was conducted on a case-control trial involving 60 children (29 boys, 31 girls) as part of a public education initiative hosted on the web-based platform "Hand in Hand Across Barriers - Public Education Platform" (Facebook).

DETAILED DESCRIPTION:
The program consisted of short, age-appropriate animated narratives reflecting three Home-FAST domains: (1) Home Environment and Furniture, (2) Capability in Activities of Daily Living, and (3) Use of Devices. Pre- and post-intervention assessments included knowledge quizzes and caregiver-supported completion of the 74-item pictorial HSSAT v.5 checklist.

ELIGIBILITY:
Inclusion Criteria:

* full time students

Exclusion Criteria:

* know neurological disorder

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: students who were studying in primary school
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2025-04-02 (Actual); Study Completion 2025-04-02 (Actual)

PRIMARY OUTCOMES:
HSSAT (v.5) | 20mins
  The HSSAT (v.5) checklist examines and provides solutions for 10 specific areas of the home: Entrance to Front Door and Front Yard (1), Entrance to Back/Side Door (2), Hallway or Foyer (3), Living Room (4), Kitchen (5), Bedroom (6), Bathroom (7), Staircases (8), Laundry Room/Basement (9), Garage (10).

CONTACTS AND LOCATIONS:
Overall Officials: Frank Lai, PhD, Principal Investigator — Northumbria University
Locations (1):
- Northumbria University, Newcastle, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
This will be shared upon reasonable request with academic purposes